CLINICAL TRIAL: NCT04694950
Title: Postoperative Recovery and Comfort After Urologic Robotic Surgery: A Feasibility Study
Brief Title: Postoperative Recovery and Comfort in Patients Undergoing Urologic Robotic Surgery
Status: Completed | Type: Observational
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Martin Holmberg, Principal investigator, Linkoeping University
Other Study IDs: 210101
Record Dates: First submitted 2020-12-29; First posted 2021-01-05 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Quality of Recovery; Urology; Pain; PONV; Postoperative Complications; Laparoscopic
MeSH Terms: conditions — Pain; Postoperative Nausea and Vomiting; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group feasibility: Adults undergoing elective urologic laparoscopic robotic surgery.
  Interventions: Procedure: Usual care

INTERVENTIONS:
Procedure: Usual care — Intravenous morphine according to clinician´s discretion.

SUMMARY:
Previously published studies show that adding intrathecal morphine to general anesthesia can reduce the postoperative pain and length of stay (LOS) in varies types of surgery. A recent meta-analysis showed that the addition of intrathecal morphine at doses below 500µg did not increase the risk of respiratory depression compared with a control group receiving intravenous opioids. Epidural analgesia is uncommonly used for robot-assisted laparoscopic procedures due to the limited surgical trauma. In addition, the risks associated with the epidural itself such as infection and spinal hematoma are thought to outweigh its possible benefits for these procedures.

At Linkoping University Hospital a combination of general anesthesia and intrathecal morphine in robot-assisted laparoscopic radical prostatectomy and in robotic-assisted laparoscopic cystectomy is now routinely used in order to improve postoperative recovery. However whether this approach is beneficial in other types of robotic-assisted urological procedures is unknown.

Therefore the investigators aim to conduct a feasibility study for the use of intrathecal morphine combined with general anaesthesia in adult patients undergoing elective urologic laparoscopic robot-assisted surgery at Linkoping University Hospital. The investigators will include 30 patients in the study. The specific aims are to investigate the feasibility and sensitivity of Quality of Recovery 15 (QoR15), as an outcome tool measuring postoperative well-being in this patient cohort.

The investigators will also investigate the feasibility of other outcome measures such as postoperative pain, post-anesthesia care unit LOS, occurrence of pruritus and hospital LOS.

For planning of the timeframe of the future interventional study the investigators will use this feasibility study to examine the inclusion rate of study patients.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective urologic robotic assisted laparoscopic surgery in Linkoping University Hospital

Exclusion Criteria:

* Age <18
* Not expected to comprehend the written or verbal study information
* Patient planned for robotic assisted laparoscoic prostatectomy or robotic assisted laparoscopic cystectomy
* Acute surgery
* ASA class >3
* Major surgery on another organ planned at the same operation
* Patient planned for a neuraxial blockade in addition to general anaesthesia.
* Study personal not available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult population undergoing elective urologic robotic assisted laparoscopic surgery in Linkoping University Hospital, sweden.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2021-10-19 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Recovery 15 (QoR-15) score | Preoperative, postoperative up to day 7
  Quality of Recovery 15. A total of 15 questions each answered with a value from 0 to 10. The minimum value of the QoR-15 is 0 and the maximum value is 150. A higher value means a better outcome.

SECONDARY OUTCOMES:
Postoperative pain | Up to postoperative day 3
  Measurement of pain in rest and in movement with the Numeric Rating Scale (NRS) Pain Scale. Minimum value is 0 (no pain) and maximum value is 10 (extreme pain).
PONV | Up to postoperative day 3
  Measurement of the frequency of postoperative nausea and vomiting (PONV).
Return of bowel function | Up to postoperative day 7
  Time to first passing of flatus and first passing of stool.
Postoperative complications | Up to postoperative day 30
  Using the Clavien-Dindo Classification
Length of hospital stay | Up to 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Chew, MD PhD, Study Director — Linkoeping University
Locations (1):
- Linkoping University Hospital, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No